CLINICAL TRIAL: NCT00090298
Title: A Multicenter, Randomized, Double-Blind Study to Evaluate the Lipid-Altering Efficacy and Safety of the Ezetimibe/Simvastatin Combination Tablet Versus Rosuvastatin in Patients With Primary Hypercholesterolemia
Brief Title: Study to Evaluate the Cholesterol Lowering Effects of Two Marketed Drugs in Patients With Elevated Cholesterol Levels (0653A-058)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-058; 2004_001
Record Dates: First submitted 2004-08-25; First posted 2004-08-30 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653A, ezetimibe (+) simvastatin
Drug: Comparator: Rosuvastatin

SUMMARY:
A 10-week study to compare the reduction in cholesterol following treatment with two different marketed drugs in patients with hypercholesterolemia.

DETAILED DESCRIPTION:
The duration of treatment is 6 weeks.

ELIGIBILITY:
Men and women aged 18 to 69 years, with elevated cholesterol levels may be eligible to participate in a research study to assess the efficacy and safety of two marketed drugs.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2815 (Actual)
Dates: Start 2004-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
LDL-C lowering efficacy after 6 weeks.

SECONDARY OUTCOMES:
Safety;changes in TC, non-HDL-C, TG, HDL-C, Apo B, LDL-C/HCL-C ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Catapano AL, Davidson MH, Ballantyne CM, Brady WE, Gazzara RA, Tomassini JE, Tershakovec AM. Lipid-altering efficacy of the ezetimibe/simvastatin single tablet versus rosuvastatin in hypercholesterolemic patients. Curr Med Res Opin. 2006 Oct;22(10):2041-53. doi: 10.1185/030079906X132721. PMID 17022864